CLINICAL TRIAL: NCT03690102
Title: The Effect of Telephone Assistance on the Quality of Cardiopulmonary Resuscitation and Use of Automated External Defibrillator.
Brief Title: The Effect of T-CPR on the Quality of CPR and AED Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Collaborators: TrygFonden, Denmark (Industry); Emergency Medical Services, Capital Region, Denmark (Other Government); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Kristine Elisabeth Eberhard, Researcher, medical student, Copenhagen Academy for Medical Education and Simulation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CAMES/AkutBeredskabet_2018_001
Record Dates: First submitted 2018-09-26; First posted 2018-10-01 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Basic Cardiac Life Support; Cardiopulmonary Resuscitation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
  Participants are randomized to one of three groups (stratified for course type, using computer-generated lists with variable block sizes):
  Participants are given a cardiac arrest scenario test either before or after a European Resuscitation Council standardized basic life support course. Two of the groups receive instructions in cardiopulmonary resuscitation from a dispatcher when they call the Emergency Medical Services.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No BLS course. With T-CPR. (Experimental): The participant is presented for a cardiac arrest scenario before attending the ERC standardized BLS course.
  During the scenario test, the participant will receive T-CPR.
  Interventions: Other: T-CPR
- With BLS course. No T-CPR. (Experimental): The participant is presented for a cardiac arrest scenario after completion of the ERC standardized BLS course.
  During the scenario test, the participant will not receive T-CPR.
  Interventions: Other: ERC standardized BLS course
- With BLS course. With T-CPR. (Experimental): The participant is presented for a cardiac arrest scenario after completion of the ERC standardized BLS course.
  During the scenario test, the participant will receive T-CPR.
  Interventions: Other: T-CPR; Other: ERC standardized BLS course

INTERVENTIONS:
Other: T-CPR — Participants receive telephone instructions in cardiopulmonary resuscitation (T-CPR) from the Emergency Medical Services in Copenhagen during the cardiac arrest scenario test.
  Arms: No BLS course. With T-CPR.; With BLS course. With T-CPR.
Other: ERC standardized BLS course — Participants will receive and complete the standardized course in basic life support (BLS) from European Resuscitation Council (ERC).
  Arms: With BLS course. No T-CPR.; With BLS course. With T-CPR.

SUMMARY:
The purpose of the study is to examine the effect of telephone assistance and standardized basic life support courses on the quality of cardiopulmonary resuscitation (CPR) and the use of automated external defibrillator (AED).

The investigators hypothesize that bystanders can provide compressions in correct frequency and use an AED correctly as well as safely from telephone instructions but that correct and successful ventilations including correct open airway require training on a course.

DETAILED DESCRIPTION:
The study aims at answering the following research questions:

1. How is the quality of CPR and use of AED when performed by an inexperienced bystander who receives telephone assistance compared to the quality when performed by a trained bystander, who has passed a standardized European Resuscitation Council (ERC) course in basic life support (BLS) but does not receive telephone assistance?
2. How is the quality of CPR and use of AED when performed by a trained bystander who has passed a standardized ERC course in BLS and who receives telephone assistance compared to the quality when performed by a trained bystander who does not receive telephone assistance?

The questions are sought answered through simulated cardiac arrest scenarios in non-classroom settings.

Participants are recruited from ERC courses in BLS.

Participants are randomised to one of three groups (stratified for course type using computer-generated randomisation lists with blocks of variable sizes):

1. Cardiac arrest scenario test before BLS course with telephone-assistance.
2. Cardiac arrest scenario test after BLS course, no telephone-assistance.
3. Cardiac arrest scenario test after BLS course with telephone-assistance.

ELIGIBILITY:
Inclusion Criteria:

* Participant at a European Resuscitation Council standardized basic life support course. Participants are enrolled from courses for university students, courses for elderly and courses for recruits in the Danish Emergency Management Agency.

Exclusion Criteria:

* Basic life support course within the last two years.
* Healthcare professional or background as healthcare professional.
* Instructor in basic life support or first aid.
* Lifeguard or background as lifeguard.
* Does not want to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2020-08-23 (Actual); Study Completion 2020-08-23 (Actual)

PRIMARY OUTCOMES:
Compression depth | 8 minutes
  Keeps a compression depth as recommended by International Liaison Committee on Resuscitation (ILCOR) (5-6 cm) on at least 50 % of compressions (yes/no). Measured by advanced manikin.
Compression rate | 8 minutes
  Rescuer keeps a compression rate of approximately 100-120 compressions per min. throughout the CPR (yes/no). Measured by advanced manikin.
Shock delivered | 8 minutes
  Shock delivered with AED (yes/no). Assessed by ERC instructor.

SECONDARY OUTCOMES:
Hands-of time | 8 minutes
  Relevant actions of resuscitation within more than 75 % of the test time (yes/no). Measured as no flow time by advanced manikin.
Responsiveness | 8 minutes
  Shakes AND shouts (yes/no). Assessed by ERC instructor.
Open airway | 8 minutes
  Opens or correctly tries to open mouth (chin lift OR jaw thrust) (yes/no). Assessed by ERC instructor.
Assess breathing | 8 minutes
  Looks, listens AND feels for normal breathing (yes/no). Assessed by ERC instructor.
Recoil/lean | 8 minutes
  Full rise on at least 50 % of all compressions (yes/no). Measured by advanced manikin.
Rescue breaths | 8 minutes
  More than 400 mL for at least 50 % of all ventilations (yes/no). Measured by advanced manikin.
Ratio | 8 minutes
  Acceptable range 28-32:2 (yes/no). Assessed by ERC instructor.
Activate AED | 8 minutes
  Activates AED immediately upon arrival (yes/no). Assessed by ERC instructor.
Attachment of AED pads | 8 minutes
  Correct attachment of AED pads according to the picture in protocol (yes/no). Assessed by ERC instructor.
Stand clear | 8 minutes
  Ensures safety by looking around and verbally announcing delivery of shock (yes/no). Assessed by ERC instructor.
Compression depth 2 | 8 minutes
  Percentage of compressions with a depth within the recommendations from ILCOR (5-6 cm) (%). Measured by advanced manikin.
Compression rate 2 | 8 minutes
  Average rate of compressions (compressions/minute). Measured by advanced manikin.
Rescue breaths 2 | 8 minutes
  Percentage of ventilations with more than 400 mL (%). Measured by advanced manikin.
Time to first compression | 8 minutes
  Time from scenario start to first compression. Assessed by ERC instructor.
Hand placement | 8 minutes
  Correct hand placement in at least 50 % of compressions (yes/no). Measured by advanced manikin.

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Lippert, Study Director — Emergency Medical Services, Capital Region, Denmark; Doris Oestergaard, Study Director — Copenhagen Academy for Medical Education and Simulation
Locations (1):
- Student2Student, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No